CLINICAL TRIAL: NCT04169763
Title: A Phase I Study of Nelfinavir and Cisplatin Chemotherapy Concurrent With Pelvic Radiation for Locally Advanced Vulvar Cancer Not Amenable to Surgical Resection
Brief Title: Nelfinavir, Cisplatin, and External Beam Radiation Therapy for the Treatment of Locally Advanced Vulvar Cancer That Cannot Be Removed by Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0629; NCI-2019-07570 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0629 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Stage II Vulvar Cancer AJCC v8; Stage III Vulvar Cancer AJCC v8; Stage IIIA Vulvar Cancer AJCC v8; Stage IIIB Vulvar Cancer AJCC v8; Stage IIIC Vulvar Cancer AJCC v8; Stage IVA Vulvar Cancer AJCC v8
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiation; Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (nelfinavir, cisplatin, EBRT) (Experimental): Patients receive nelfinavir PO BID for up to 8 weeks. Starting week 2, patients also receive cisplatin IV over 60-90 minutes once weekly during weeks 2-8. Patients undergo EBRT for 5 consecutive days between weeks 2-8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Radiation: External Beam Radiation Therapy; Drug: Nelfinavir

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone''s Chloride; Peyrone''s Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
Drug: Nelfinavir — Given PO

SUMMARY:
This phase I trial studies the side effects and best dose of nelfinavir when given together with cisplatin and external beam radiation therapy in treating patients with vulvar cancer that has spread to nearby tissue or lymph nodes (locally advanced) and cannot be removed by surgery. Nelfinavir is an antiviral drug normally used to treat human immunodeficiency virus (HIV). Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy beams to kill tumor cells and shrink tumors. Giving nelfinavir, cisplatin, and external beam radiation therapy may work better than giving only cisplatin and external beam radiation therapy in treating patients with vulvar cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and dose limiting toxicities of nelfinavir in combination with cisplatin plus inguinal +/-pelvic radiation therapy for treatment of patients with unresectable T2-4, N0-3 vulvar carcinoma.

II. To determine the recommended phase II dose of nelfinavir combined with chemoradiotherapy.

SECONDARY OBJECTIVES:

I. To determine recurrence site (local/distant), progression-free survival and overall survival.

II. To determine the levels of Akt activity (and downstream effectors such as pGSK3, pEBP1) and p16INK4A in addition to the presence of human papilloma virus (HPV) 16 and 18, and E6/E7 ribonucleic acid (RNA) in vulvar biopsy specimens of patients at up to two(2) different time points (1. pre nelfinavir, pre-radiation, 2. while on nelfinavir, pre-radiation).

OUTLINE:

Patients receive nelfinavir orally (PO) twice daily (BID) for up to 8 weeks. Starting week 2, patients also receive cisplatin intravenously (IV) over 60-90 minutes once weekly during weeks 2-8. Patients undergo external beam radiation therapy (EBRT) for 5 consecutive days between weeks 2-8. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* All patients with primary, previously untreated, histologically confirmed invasive carcinoma of the vulva (any cell type) not amenable to surgical excision. Clinical stages T2-T4, N0-3, M0. Hematoxylin & eosin (H & E) stained slide showing documentation of the primary invasive cancer is required. All specimens of primary tumor require documentation of type
* Absolute neutrophil count (ANC) >= 1,500/microliter (performed within 28 days from signing consent form)
* Platelet count >= 100,000/microliter (performed within 28 days from signing consent form)
* Creatinine < 2.0 mg/dL (performed within 28 days from signing consent form)
* Total bilirubin =< 1.5 times normal (performed within 28 days from signing consent form)
* Glutamic-oxaloacetic transaminase (SGOT) =< 3 times normal (performed within 28 days from signing consent form)
* Patients with an Eastern Cooperative Oncology Group/Gynecologic Oncology Group (ECOG/GOG) performance status of 0, 1, or 2
* Patients with ureteral obstruction must be treated with stent or nephrostomy tube
* Patients must be consented within twelve (12) weeks of diagnosis or must be restaged
* Patients of childbearing potential must use an effective form of birth control. "Patients receiving oral contraceptives should be instructed that alternate or additional contraceptive measures should be used during therapy with VIRACEPT."
* Confirmed seronegative HIV status within 3 months of signing consent
* Patients must have signed an approved informed consent and authorization permitting release of personal health information

Exclusion Criteria:

* Patients with stage T1N0 disease
* Patients who have known metastases to other organs outside the radiation field at the time of the original clinical and surgical staging
* Patients who have received previous pelvic or abdominal radiation, cytotoxic chemotherapy, or previous therapy of any kind for this malignancy
* Patients with septicemia or severe infection
* Patients who have circumstances that will not permit completion of this study or the required follow-up
* Patients who are pregnant at the time of diagnosis and do not wish pregnancy termination prior to initiation of treatment
* Patients with renal abnormalities, such as pelvic kidney, horseshoe kidney, or renal transplantation, that would require modification of radiation fields
* Patients with other concomitant malignancies (with the exception of non-melanoma skin cancer), who had (or have) any evidence of other cancer present within the last 5 years
* Patients with gastrointestinal (GI) tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for intravenous (IV) alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis)
* Patients with poorly controlled diabetes mellitus despite medication
* Patients taking anti-arrhythmic agents such as amiodarone, quinidine, rifampin, ergot derivatives such as ergotamine, St John's wort, human menopausal gonadotropin (HMG)-CoA reductase inhibitors such as lovastatin, neuroleptic such as pimozide, sedatives such as midazolam and triazolam among other CYP3A4 and CYP2C19 substrates
* Patients with phenylketonuria
* Patients with estimated glomerular filtration rate (eGFR) < 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of nelfinavir | 1 year
  Defined as the dose for which the isotonic estimate of the dose limiting toxicity (DLT) rate is closest to the target DLT rate of 30%. If there are ties, the higher dose will be chosen as the RP2D when the isotonic estimate is lower than 30%, and the lower dose will be chosen when the isotonic estimate is greater than or equal to 30%.
Incidence of adverse events | 1 year
  Results from the dose escalation phase of study will be summarized by a tabulation of the number of patients treated and the number who experience a DLT at each dose level tested. Comprehensive safety data on all toxicities will be tabulated by type, grade, duration, attribution to treatment, and administered dose level. A patient level summary by worst grade toxicity will be included. Laboratory data and concomitant medications associated with episodes of toxicity will be summarized. Will also report the number of patients who discontinue therapy and the reasons for discontinuation.

SECONDARY OUTCOMES:
Progression-free survival | 1 year
  Will be estimated using the product-limit method developed by Kaplan and Meier. Will report rates at specific times (e.g., at 6 and 12 months) and medians, if attained, with corresponding 95% confidence interval.
Overall survival | 1 year
  Will be estimated using the product-limit method developed by Kaplan and Meier. Will report rates at specific times (e.g., at 6 and 12 months) and medians, if attained, with corresponding 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Lilie L Lin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Related Info — http://www.mdanderson.org